CLINICAL TRIAL: NCT00733460
Title: A Phase I Study to Evaluate the Safety, Biodistribution and Radiation Dosimetry of BFPET as a Potential Myocardial Perfusion Imaging (MPI) Agent for PET
Brief Title: A Phase I Study to Evaluate BFPET as a Potential Myocardial Perfusion Imaging(MPI) Agent for PET
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fluoropharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BFPET P-01
Record Dates: First submitted 2008-08-12; First posted 2008-08-13 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2013-06

CONDITIONS: Coronary Artery Disease
Keywords: BFPET; Coronary Artery Disease; Myocardial Perfusion Imaging; Radiation Dosimetry
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BF-PET (Experimental)
  Interventions: Drug: BFPET

INTERVENTIONS:
Drug: BFPET

SUMMARY:
Safety and dosimetry of BFPET™ will be evaluated in healthy volunteers and Coronary Artery Disease (CAD) patients , male or female and of age ranging between 20-80 years old.

DETAILED DESCRIPTION:
Study Procedures:

Visit 1: Screening - Eligibility determination

Visit 2 (within 14 days post screening): Injection of BFPET™ and PET Imaging

Visit 3 (within 24-48 hours post dose): Follow-up Visit

ELIGIBILITY:
NORMAL HEALTHY VOLUNTEERS Inclusion Criteria

1. Subject must provide written informed consent prior to any study related procedures;
2. Subject must be ≥ 20 and ≤ 80 years of age;
3. Subject must have a serum creatinine within the investigational site's normal range.
4. Subject must have liver function tests < 1.5 times the investigational site's normal range.
5. Subject must have a hematocrit level within 5% of the investigational site's normal range.

Exclusion Criteria:

1. Any clinically significant acute or unstable physical or psychological disease based on medical history or screening physical examination;
2. Any clinically significant abnormality in the screening laboratory tests or ECG;
3. Any exposure to any investigational drugs within four (4) weeks prior to Visit 1;
4. Any exposure to investigational radiopharmaceuticals within four (4) weeks prior to the date of Visit 1;
5. Any new prescription medications within four (4) weeks of Visit 1;
6. Subject has a Positive (+) Serum Pregnancy Test, or the possibility of pregnancy cannot be ruled out prior to dosing or is breast-feeding. There are standard pregnancy procedures for use of radiopharmaceuticals in research at MGH.
7. Subject has experienced any allergic reaction to similar radiofluorinated compounds or agents.

CORONARY ARTERY DISEASE (CAD) SUBJECTS

Inclusion Criteria:

1. Subjects must provide written informed consent prior to any study related procedures;
2. Subjects must be ≥ 20 and ≤ 80 years of age;
3. Subjects must have history of CAD documented by an abnormal stress myocardial perfusion imaging (MPI) study and cardiac catheterization within 6 months of the BFPET studyExclusion Criteria

Exclusion Criteria:

1. Subject has a Positive (+) Serum and/or Urine Pregnancy Test or is lactating, or the possibility of pregnancy cannot be ruled out prior to dosing;
2. Any clinically significant acute or unstable physical or psychological disease judged by the investigators based on medical history or screening physical examination;
3. Coronary artery bypass graft (CABG) within 6 months;
4. Percutaneous coronary intervention (PCI), with stent placement within six months;
5. Blood pressure over 180/100;
6. Acute changes in ECG;
7. Recent (within 3 months) cardiac arrest, unstable angina, myocardial infarction, cerebro-vascular accident (CVA), any general anesthesia procedure, any surgical procedures;
8. Any implanted pacemaker or defibrillator use within the last three months;
9. Inability to remain in camera for approximately 60 minutes (Smokers and COPD are included as long as they can breath in PET camera and not taking O2 through nasal canula);
10. History of Diabetes Mellitus;
11. Serum creatinine > 2 mg/dL;
12. All cancer patients;
13. Body Mass Index (BMI) is over 35;
14. Any exposure to any investigational drugs or medical device within four (4) weeks prior to imaging study;
15. Any exposure to radiopharmaceuticals within four (4) weeks prior to the date of imaging study;

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-03; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure. Safety Biodistribution Radiation dosimetry | pre-dose, post-dose 0, 1, 5, 15, 30, 60 and 90 minutes, 2 hours, 24-48 hours post-dose and 7 days post-dose.
  Change in vital signs, physical examination, ECG measured within 14 days of screening, immediate pre-dose, post-dose and 24-48 hours post-dose.
  Change in 12-lead Electrocardiogram measured within 14 days of screening, immediate pre-dose, post-dose and 24-48 hours post-dose.
  Change in 24-hour Holter (initiated 2 hours pre-dose, continuous for 24 hours, time stop recorded.
  Change in dosimetry sampling (blood and urine)blood measured at time 0 (immediately following injection), 1,5, 15, 30, 60, 90 minutes.
  Adverse event assessment immediate post dose, 24-48 hours and 7 days post-dose.

SECONDARY OUTCOMES:
Performance characteristics of BFPET as a PET tracer for myocardial imaging. | 30, 60, 120, and 240 seconds.
  Whole body imaging measures radiation dosimetry at rest and under pharmacologic stress

CONTACTS AND LOCATIONS:
Overall Officials: Henry Gewirtz, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States